CLINICAL TRIAL: NCT06574347
Title: A Phase II Study of Vebreltinib Plus PLB1004 as the First-line Therapy for Patients With EGFRm+/MET+ Locally Advanced or Metastatic Non-small Cell Lung Cancer.
Brief Title: Vebreltinib Plus PLB1004 as the First-line Therapy for Patients With EGFRm+/MET+ Locally Advanced or Metastatic NSCLC.
Acronym: KYLIN-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Avistone Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PLB1001/PLB1004-NSCLC-II-02
Record Dates: First submitted 2024-08-25; First posted 2024-08-27 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2024-08

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: NSCLC; Lung Cancer; MET Amplification; EGFR L858R; EGFR Exon 19 Deletion; EGFR
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vebreltinib 150mg BID+PLB1004 80mg QD (Experimental): Subjects will receive Vebreltinib 150mg orally twice per day (BID) + PLB1004 80mg orally once per day (QD),21day cycles until disease progression, death, adverse event (AE) leading to discontinuation or withdrawal of consent.
  Interventions: Drug: Vebreltinib; Drug: PLB1004
- Osimertinib 80mg QD (Active Comparator): Subjects will receive Osimertinib 80mg orally once per day (QD),21day cycles until disease progression, death, adverse event (AE) leading to discontinuation or withdrawal of consent.
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Vebreltinib — Subjects will receive Vebreltinib orally twice per day (BID).
  Other Names: Bozitinib; PLB1001
  Arms: Vebreltinib 150mg BID+PLB1004 80mg QD
Drug: Osimertinib — Subjects will receive Osimertinib 80mg orally once per day (QD).
  Other Names: AZD9291
  Arms: Osimertinib 80mg QD
Drug: PLB1004 — Subjects will receive PLB1004 80mg orally once per day (QD).
  Other Names: Andamertinib
  Arms: Vebreltinib 150mg BID+PLB1004 80mg QD

SUMMARY:
Efficacy and Safety Evaluation of Vebreltinib Plus PLB1004 as the First-line Therapy for Patients With EGFRm+/MET+ Locally Advanced or Metastatic NSCLC.

DETAILED DESCRIPTION:
A Multicenter,Randomized,open-label,Phase II Study to Evaluate the Efficacy and Safety of Vebreltinib Plus PLB1004 as the First-line Therapy for Patients with EGFRm+(exon 19 deletion or exon 21 L858R)/MET+ Locally Advanced or Metastatic Non-small Cell Lung Cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to sign a written informed consent document.
2. Aged at least 18 years old.
3. Histologically or cytologically confirmed locally advanced or metastatic NSCLC (stage IIIB~IV).
4. Patients with previously untreated, EGFRm-positive (exon 19 deletion or L858R) and MET overexpression (IHC 3+) .
5. At least one measurable lesion as defined by RECIST V1.1.
6. ECOG performance status 0 to 1.

Exclusion Criteria:

1. There are mutations of ALK or ROS1.
2. Have symptomatic and neurologically unstable central nervous system (CNS) metastases or CNS disease that requires increased steroid doses for control.
3. Pregnant or nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
The objective response rate of the tumor (ORR) | 2 Years
  The incidence of confirmed complete response or partial response.

SECONDARY OUTCOMES:
The disease control rate (DCR) | 2 Years
  The incidence of complete response, partial response and stable disease.
Duration of Response (DoR) | 2 Years
  The duration between the date the criteria for complete response or partial response was first measured (first record shall prevail) and the date of disease recurrence or progression as objectively recorded.
Progression-free survival (PFS) | 2 Years
  Progression-free survival (PFS) using Investigator assessment as defined by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1).
Time to Response (TTR) | 2 Years
  The period from the date of randomization to the date when the criteria for complete response or partial response was first measured (first record shall prevail).
Incidence of Treatment-Emergent Adverse Events | 2 Years
  Incidence of Treatment-Emergent Adverse Events (TEAEs),A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Yi long Wu, MD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China